CLINICAL TRIAL: NCT01270321
Title: A 3-Arm Randomized Phase II Trial Evaluating Single Agent and Combined Efficacy of Pasireotide and Everolimus in Adult Patients With Radioiodine-Refractory Differentiated and Medullary Thyroid Cancer
Brief Title: Pasireotide & Everolimus in Adult Patients With Radioiodine-Refractory Differentiated & Medullary Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Taofeek K. Owonikoko, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00041909; WCI1777-09 (Other: Other)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2020-08-25 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Everolimus; pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Everolimus alone) (Experimental): CURRENTLY CLOSED TO ACCRUAL--Everolimus alone followed by Everolimus + Pasireotide at the time of progression
  Interventions: Drug: Everolimus
- Arm B (Pasireotide alone) (Experimental): CURRENTLY CLOSED TO ACCRUAL--Pasireotide alone followed by Everolimus + Pasireotide at the time of progression
  Interventions: Drug: Pasireotide
- Arm C (Everolimus + Pasireotide) (Experimental): CURRENTLY CLOSED TO ACCRUAL
  Interventions: Drug: Everolimus and Pasireotide

INTERVENTIONS:
Drug: Everolimus — Everolimus 10 mg daily continuously (switch to 2-drug combination at progression if no intolerable toxicity)
  Other Names: Afinitor; RAD001
  Arms: Arm A (Everolimus alone)
Drug: Pasireotide — Pasireotide 1200 mcg bid for 4 weeks followed by Pasireotide long acting release (LAR) 60 mg i.m. once every 4 weeks
  Other Names: SOM230
  Arms: Arm B (Pasireotide alone)
Drug: Everolimus and Pasireotide — Everolimus 10 mg daily continuously together with Pasireotide 1200 mcg bid for 4 weeks followed by Pasireotide long acting release (LAR) 60 mg i.m. once every 4 weeks
  Other Names: Afinitor; SOM230
  Arms: Arm C (Everolimus + Pasireotide)

SUMMARY:
The purpose of this study is to determine the effectiveness of two anticancer drugs, everolimus and pasireotide, in patients with thyroid cancer when the cancer is no longer responding to treatment with radioiodine or where it is deemed unsafe for the patient to receive additional radioiodine treatment. The investigators also want to establish the best manner of taking the two medications when used together to treat thyroid cancer. In particular, the investigators want to know if it is better to give both at the same time or add a second medication after the first one has stopped working.

This study will also look at specific substances called biomarkers in your blood, and in the tumor tissue which are involved in the growth of tumor cells, and determine if the levels of these biomarkers are related to your response to treatment or development of side effects.

Everolimus, also known by the brand name, Afinitor, is a biologic drug approved by the Food and Drug Administration (FDA) for the treatment of kidney cancer. It works by preventing cancer cells from multiplying and it also makes them more likely to die from the treatment.

Pasireotide also known by the name, SOM230 is a new medication that is not yet approved by the FDA for the treatment of cancer. It is a newer form of a drug called octreotide, which is approved for the treatment of cancer arising from endocrine organs. Pasireotide works by binding to a protein called somatostatin receptor, which is expressed in many tissues throughout the body including thyroid cancer cells. Pasireotide prevents the action of somatostatin by binding to these receptors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic confirmation of thyroid cancer (papillary, follicular, medullary); histologic variants such as Hurthle and tall cell variants are allowed.
2. Biochemical or radiologic documentation of disease progression within the last 12 months prior to enrollment.
3. Presence of at least one site of measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
4. Patient must have radioiodine refractory disease as defined by one or more of the following conditions:

   * All cases of medullary thyroid carcinoma.
   * No iodine-uptake on a post- radioactive iodine treatment scan (in presence of low iodine diet and thyroid stimulating hormone (TSH) suppression) in an anatomically defined lesion that qualifies as target lesion by RECIST criteria.

   OR

   • If there is demonstrable iodine-uptake: the last radioiodine therapy of (≥ 100 mCi) was given within the last 16 months OR if given more than 16 months before enrollment, there is evidence of disease progression after each of the last two radioiodine treatment performed within 16 months of each other (each dose should be ≥ 100mCi).

   OR
   * If the patient has received the maximum cumulative life time dose of radioactive iodine treatments of at least 600 mCi.
   * If the patient declines or is intolerant of radioiodine therapy or if with progressive disease that is, in the opinion of the treating physician, likely to benefit from biologic therapy rather than further iodine therapy e.g. patient with heavy burden of disease
5. Age ≥ 18 years.
6. Minimum of four weeks since any major surgery or since completion of radiation (patients should have adequately recovered from the acute toxicities of any prior therapy).
7. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
8. Life expectancy of at least 6 months.
9. Adequate bone marrow function as shown by: absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L, platelets ≥ 100 x 10⁹/L, Hgb > 9 g/dL.
10. Adequate liver function as shown by: serum bilirubin ≤ 1.5 x upper limit of normal (ULN), and serum transaminases activity ≤ 3 x ULN, with the exception of serum transaminases (< 5 x ULN) if the patient has liver metastases.
11. Adequate renal function as shown by serum creatinine ≤ 1.5 x ULN or glomerular filtration rate (GFR) of 60cc/ml using the formula of Cockroft and Gault.
12. Fasting serum cholesterol ≤ 300 mg/dL OR ≤ 7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN. NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
13. Women of childbearing potential must have a negative serum pregnancy test within 14 days of the administration of the first study treatment. Women must not be lactating. Both men and women of childbearing potential must be advised of the importance of using effective birth control measures during the course of the study.
14. Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.
15. International normalized ratio (INR) and prothrombin time (PTT) ≤ 1.5 x ULN. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of low molecular weight [LMW] heparin for > 2 weeks at time of randomization.)

Exclusion Criteria:

1. Prior treatment with not more than 1 systemic agent.
2. Patients who have undergone major surgery within 4 weeks prior to study enrollment (tracheotomy, feeding tube or vascular access catheter placement and interventional procedures such as bronchoscopy, upper GI endoscopy or colonoscopy are not considered major surgery).
3. Chronic treatment with systemic steroids or another immunosuppressive agent.
4. Patients should not receive immunization with attenuated live vaccines during study period or within 1 week of study entry.
5. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases.
6. Patients with prior or concurrent malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years.
7. Patients with uncontrolled diabetes mellitus or a fasting plasma glucose > 1.5 ULN. Note: At the principal investigator's discretion, non-eligible patients can be re-screened after adequate medical therapy has been instituted.
8. Patients with symptomatic cholelithiasis (asymptomatic gall stone discovered on screening US should be reviewed by the PI but will not lead to automatic exclusion).
9. Liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C):

   * History of liver disease, such as cirrhosis or chronic active hepatitis B and C.
   * Presence of Hepatitis B surface antigen (HbsAg).
   * Presence of Hepatitis C antibody test (anti-HCV).
10. Patients who have congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block or a history of acute myocardial infarction within the six months preceding enrollment.
11. QT related exclusion criteria:

    * QT corrected Fridericia's method (QTcF) at screening > 470 msec.
    * History of syncope or family history of idiopathic sudden death.
    * Sustained or clinically significant cardiac arrhythmias.
    * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade atrioventricular (AV) block.
    * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure.
    * Concomitant medication(s) known to increase the QT interval.
12. Patients with the presence of active or suspected acute or chronic uncontrolled infection or with a history of immunocompromise, including a positive HIV test result (ELISA and Western blot).
13. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

    * Severely impaired lung function (as defined as spirometry and diffusing capacity of lung for carbon monoxide [DLCO] that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air).
    * Any active (acute or chronic) or uncontrolled infection/disorders.
    * Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy.
    * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (everolimus).
    * Patients who have a history of alcohol or drug abuse in the 6 month period prior to receiving treatment with pasireotide or RAD001.
    * History of, or current alcohol misuse/abuse within the past 12 months.
    * Acute or chronic pancreatitis.
14. Women who are pregnant or breast feeding, or women/men of reproductive potential who are not using and unwilling to practice an effective method of birth control. (Women of childbearing potential [WOCBP] must have a negative serum pregnancy test within 7 days prior to administration of pasireotide and RAD001.)
15. Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment.
16. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients.
17. Known hypersensitivity to somatostatin analogues or any component of the pasireotide or octreotide LAR formulations.
18. History of noncompliance to medical regimens.
19. Patients unwilling to or unable to comply with the protocol.
20. Patients taking medications known to be strong cytochrome P450, family 3, subfamily A (CYP3A) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-11; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taofeek Owonikoko, MD, PhD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled between 11/17/2010 and 1/2/2019 at Winship Cancer Institute of Emory University
Period: Overall Study
Arm/Group | Arm A (Everolimus Alone) | Arm B (Pasireotide Alone) | Arm C (Everolimus + Pasireotide)
Started | 19 | 11 | 12
Completed | 9 | 1 | 3
Not Completed | 10 | 10 | 9
Not completed — Death | 3 | 1 | 4
Not completed — Adverse Event | 7 | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Everolimus Alone) | Arm B (Pasireotide Alone) | Arm C (Everolimus + Pasireotide) | Total
Number analyzed (Participants) | 19 | 11 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 4 | 7
  >=65 years | 17 | 10 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] — The measure of dispersion data are not available. All efforts were made to obtain these data from the PI and the study documentation.
  Years | 66.95 (NA) — There is no standard deviation for this trial | 64.73 (NA) — There is no standard deviation for this trial | 58.83 (NA) — There is no standard deviation for this trial | 60.75 (NA) — There is no standard deviation for this trial
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 5 | 15
  Male | 12 | 8 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 18 | 9 | 9 | 36
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 0 | 6
  White | 15 | 5 | 11 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: Participants]
  United States | 19 | 11 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Per Responsive Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0)
Description: Number of participants with response per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Everolimus Alone): CURRENTLY CLOSED TO ACCRUAL--Everolimus alone followed by Everolimus + Pasireotide at the time of progression
  Everolimus: Everolimus 10 mg daily continuously (switch to 2-drug combination at progression if no intolerable toxicity)
  Most frequent adverse events in >20% of patients:
  * Dry skin
  * Dysgeusia
  * Hypoalbuminemia
  * Joint Pain
  * Cough
  * Diarrhea
  * Hypercholesterolemia
  * Hypertriglceridemia
  * Hypokalemia
  * Hyponatremiapnia
  * Mucositis
  * Rash
  * Thrombocyto
- Arm B (Pasireotide Alone): CURRENTLY CLOSED TO ACCRUAL--Pasireotide alone followed by Everolimus + Pasireotide at the time of progression
  Pasireotide: Pasireotide 1200 mcg bid for 4 weeks followed by Pasireotide long acting release (LAR) 60 mg i.m. once every 4 weeks.
  Most frequent adverse events in >20% of patients:
  * Hyperbilirubinemia
  * Hypertriglyceridemia
  * Hypercholesterolemia
- Arm C (Everolimus + Pasireotide): CURRENTLY CLOSED TO ACCRUAL
  Everolimus and Pasireotide: Everolimus 10 mg daily continuously together with Pasireotide 1200 mcg bid for 4 weeks followed by Pasireotide long acting release (LAR) 60 mg i.m. once every 4 weeks.
  Most frequent adverse events in >20% of patients:
  * Hypercholesterolemia
  * Anemia
  * Headache
  * Decreased Appetite
  * Cough
  * Mucositis
  * Hyponatremia
Arm/Group | Arm A (Everolimus Alone) | Arm B (Pasireotide Alone) | Arm C (Everolimus + Pasireotide)
Number analyzed (Participants) | 19 | 11 | 12
Participants | 17 | 9 | 11

2. Secondary Outcome: Number of Participants With Progression-free Survival
Description: Time from starting treatment until disease progression as defined using Response Evaluation CriteriaIn Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or death.
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Everolimus Alone) | Arm B (Pasireotide Alone) | Arm C (Everolimus + Pasireotide)
Number analyzed (Participants) | 19 | 11 | 12
Participants | 17 | 9 | 11

ADVERSE EVENTS:
Time Frame: Adverse events collected through study completion, an average of 1 year.
Description: Any undesirable any unfavorable signs or symptom reported by the patient while on study drug .
Arm/Group | Arm A (Everolimus Alone) | Arm B (Pasireotide Alone) | Arm C (Everolimus + Pasireotide)
All-Cause Mortality (participants affected / at risk) | 3/19 | 1/11 | 4/12
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT01270321/Prot_SAP_000.pdf